CLINICAL TRIAL: NCT05824312
Title: Health-related Quality of Life of Patients With Locally Advanced Thyroid Cancer Receiving Targeted Therapy
Brief Title: HRQOL in Locally Advanced Thyroid Carcinoma
Acronym: LATCQOL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: FJCH_HNS_QOL01
Record Dates: First submitted 2023-03-28; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Thyroid Cancer; Tyrosine Kinase Inhibitor; Health Related Quality of Life
Keywords: HRQOL; thyroid cancer; targeted therapy; Tyrosine kinase inhibitor
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TKI group: patients with LATC receiving Tyrosine kinase inhibitor drugs.
  Interventions: Drug: Tyrosine kinase inhibitor drugs.
- Controlled group: patients with LATC receiving other treatment.

INTERVENTIONS:
Drug: Tyrosine kinase inhibitor drugs. — TKI drugs were used at least 8 weeks. Imaging exam would be taken every four weeks.
  Other Names: TKI treatment
  Groups: TKI group

SUMMARY:
The purpose of this study was to explore the changes of health-related quality of life (HRQOL) in patients with locally advanced thyroid cancer (LATC) receiving TKI drugs (anlotinib, lenvatinib, etc.).

DETAILED DESCRIPTION:
Surgical resection is the cornerstone of treatment for thyroid cancer. However, some patients present with locally advanced disease at the time of diagnosis, and they are not eligible for radical resection. Another patients still had the risk of recurrence after surgery, endocrine therapy and iodine-131 treatment. Tyrosine kinase inhibitors (TKI) have been proved to be effective in thyroid cancer patients. However, it was still unclear whether TKI drugs had influence on the HRQOL of LATC patients. The purpose of this study was to explore the changes of health-related quality of life (HRQOL) in patients with locally advanced thyroid cancer (LATC) receiving TKI drugs (anlotinib, lenvatinib, etc.).Participants enroll the study after informed consent, and quality of life will be assessed using quality of life questionnaires EORTC QLQ C30, and EORTC THY 47 before surgery, and 1,3,6 and 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients age (18-70 year old)
* Diagnosis of locally advanced thyroid cancer
* Patient receiving TKI drugs.

Exclusion Criteria:

* pregnancy or breastfeeding women;
* history of other malignant diseases, unstable angina, myocardial infarction, cerebral infarction or cerebral hemorrhage within 6 months; (3) patients missing questionnaires greater than 3 times.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: locally advanced thyroid cancer
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
the global status of QLQ C30 questionnaire | 1 year
  Change in global HRQOL score between baseline and at 12 months after treatment. A change of more than 10% is set as a limit for a significant change

SECONDARY OUTCOMES:
Adversed events of TKI. | 1 year
  all TKI-related adversed events during and after the treatment of TKI.
Change in fatigue score | 1 year
  Change in fatigue score between start and at 12 months after thyroid treatment. A change of more than 10% is set as a limit for a significant change.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Study Chair — FujianMedical University Cancer Hospital
Locations (1):
- Road Fuma No.420, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No